CLINICAL TRIAL: NCT06061055
Title: Comparison of VentiBroncTM Anchor With Conventional Double-lumen Endobronchial Tube in Patients With High Risk of Malposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-2023-0043
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anchor (Experimental): Patient group who are intubated with triple-cuffed double-lumen endobronchial tube (VentiBronc Anchor)
  Interventions: Device: Intubation with VentiBronc Anchor endobronchial double-lumen tube
- Shiley (Active Comparator): Patient group who are intubated with conventional double-lumen endobronchial tube (Shiley)
  Interventions: Device: conventional double-lumen intubation

INTERVENTIONS:
Device: Intubation with VentiBronc Anchor endobronchial double-lumen tube — Patients in this group are intubated with triple-cuffed double-lumen endobronchial tube (VentiBronc Anchor).
  Arms: Anchor
Device: conventional double-lumen intubation — Patients in this group are intubated with conventional double-lumen endobronchial tube (Shiley).
  Arms: Shiley

SUMMARY:
The investigators intend to compare the group using triple-cuffed endobronchial tube (VentiBroncTM Anchor) with the group using the conventional double-lumen endotracheal tube (Shiley®) in patients at high risk of malposition of the double-lumen endotracheal tube. The aim of this study is to determine if the use of VentiBroncTM Anchor increases the success rate of optimal double-lumen intubation to left main bronchus.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring left double-lumen endotracheal tube intubation for thoracic surgery.

ASA physical status classification 2-4. Female patients aged 20-85 with a height of 160cm or less and a body mass index (BMI) of 25.0 kg/m2 or higher.

Patients requiring VentiBroncTM Anchor 33Fr or Shiley® 32Fr intubation due to a left mainstem bronchus diameter of 11mm or less on chest CT.

Exclusion Criteria:

Intraluminal lesions in the left or right mainstem bronchi. History of airway surgery. Emergency surgery.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Success rate of endobronchial intubation | Immediately after double-lumen tube intubation, with flexible fiberoptic bronchoscope
  Success or failure of endobronchial intubation will be determined immediately after double-lumen tube intubation, with flexible fiberoptic bronchoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuho Lee, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim N, Oh YJ, Kim HJ, Lee K. Novel Triple-Cuff versus Conventional Double-Cuff Double-Lumen Endobronchial Tube in Patients with Risk Factors for Tube Misdirection. Yonsei Med J. 2025 Dec;66(12):866-873. doi: 10.3349/ymj.2025.0060. PMID 41287499